CLINICAL TRIAL: NCT05042869
Title: Preliminary Study Evaluating Feasibility and Acceptability of a Psychological Management Program Focused on Body Dissatisfaction in Eating Disorders. SABG : Secondary Alveolar Bone Grafting
Brief Title: Feasibility and Acceptability of a Body Dissatisfaction Program in Eating Disorders Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0551
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Eating Disorders
Keywords: Psychiatry; Acceptance and Commitment Therapy; Body dissatisfaction
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cognitive model of Eating Disorders (ED) highlights dysfunctional cognitive patterns common to the different subtypes. Body dissatisfaction, which can be defined as the negative and subjective evaluation of one's body shape, i.e., negative thoughts and emotions concerning one's body image and the origin of pathological behaviours with the aim of modifying one's weight and body shape, thus appears to be a central transdiagnostic concept in the ED. It is, moreover, described as a major factor in the development, maintenance and relapse of the various types of ED.

It is suggested that Acceptance and Commitment Therapy (ACT) may be beneficial in treating body dissatisfaction insofar as body image inflexibility appears to influence the relationship between body image appraisal and coping strategies. ACT, which aims to develop psychological flexibility, appeared to us as a promising tool to manage body dissatisfaction in ED.

The investigators therefore aim to evaluate the feasibility and acceptability of a psychological management group for body dissatisfaction (9 or 10 weekly group session), based on ACT therapy, in patients suffering from an ED.

ELIGIBILITY:
Inclusion criteria:

* Women over 16 years
* Eating disorder, according to DSM-5 criteria (all types of eating disorder are included: anorexia, bulimia, binge eating disorder, …)
* Marked body dissatisfaction
* BMI > 17.5 kg/m2

Exclusion criteria:

* Refusal to participate
* Current severe psychiatric condition other than an ED that may impair patients' ability to attend the group
* Pregnant or breastfeeding women
* Protection measure or deprivation of liberty by administrative decision

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eating Disorders patients participating in a body dissatisfaction management program
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of the body dissatisfaction program | Day 1
  Participation rate in group sessions

SECONDARY OUTCOMES:
Acceptability of the body dissatisfaction program | day 1
  Satisfaction survey
Evolution of the eating disorder symptomatology | day 1
  Eating disorder symptomatology assessed with the Eating Disorder Examination (EDE-Q). Higher scores on the global scale and
Evolution of the eating disorder symptomatology | day 1
  Eating disorder symptomatology assessed with the Eating Disorder Inventory (EDI-2). Higher scores on the global scale and subscales indicate more severe disorder.
Evolution of the body dissatisfaction level | day 1
  Level of body dissatisfaction assessed with EDE-Q body weight and shape concerns subscales. Higher scores indicate higher body dissatisfaction
Quality of life evolution | day 1
  Quality of life assessed with Eating Disorders Quality Of Life

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Guillaume, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC